CLINICAL TRIAL: NCT05002114
Title: Evaluation of a Specific Transdermal Cannabidiol Product for Chronic Musculoskeletal Joint Pain.
Acronym: CBD001
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: there were issues with the primary study material that prohibited continuation at this time
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Principal Investigator, James C. Patterson, II, MD. Ph, Clinical Director, Louisiana Addiction Research Center, Louisiana State University Health Sciences Center Shreveport
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IND_CBD_001
Record Dates: First submitted 2021-08-02; First posted 2021-08-12 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Musculoskeletal Joint Pain
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: double-blind, randomized, placebo-controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind, randomized, placebo-controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): Does not get active topical CBD. Instead, gets an identical placebo-containing topical agent.
  Interventions: Other: Placebo
- Active Group (Experimental): Does get active topic CBD.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Topical CBD cream - special formulation
  Arms: Active Group
Other: Placebo — Not the drug
  Arms: Placebo Group

SUMMARY:
Double-blind, randomized into two arms (TC and TP): patients get either topical cannabidiol or topical placebo up to three times daily. Inclusion criteria will be chronic joint pain with intent to treat or currently treated with opioids. Exclusion criteria will include current cannabis use, severe medical illness or lacking in capacity to be involved in study. TC and TP will be prescribed for use TID in predefined dosages and quantities.

DETAILED DESCRIPTION:
Introduction and Rationale

Currently, the opioid epidemic is a public health crisis. Use of opioids for chronic pain are a large component of this crisis. If alternative means can be developed to treat chronic pain that can replace the use of opioid-based treatments, this can improve clinical outcomes and quality of life.

Arthritis and musculoskeletal pain are often chronic conditions that cause significant morbidity. Historically, one study estimated that the lifetime incidence is as high as 47% for osteoarthritis over the lifespan, increasing with age and also increasing to 60% with a body mass index over than 30. In our society today with over 50% of the population suffering from obesity, this is a significant problem.

While cannabis products have been referenced for treating numerous medical issues including a number of pain-related conditions, it has only been recently that mechanisms outside the central nervous system have been recognized. There is very little published in regards to the use of cannabidiol (CBD) in the treatment of arthritic pain, and even less on the topical application of CBD products in its use in this manner. Two previous studies demonstrated the efficacy of a local/transdermal application of CBD in rodent models of arthritis. Activity at the TRPV2 receptor is one possible mechanism for this putative mechanism. Another possible interaction is at the GPR55 receptor.

The earliest known references to the medicinal properties of cannabis can be found in the "Shennong Ben Cao Jing", which describe Chinese uses of herbal remedies from as early as 2700 BC. In later compilations of this work, cannabis is described as being utilized for the treatment of pain and inflammation. Since that time, cannabis has been used world-wide both medicinally and for recreational purposes. It has only been a recent development (within the past 100 years) that public health regulations have prohibited the use of cannabis products.

However, problems do exist with the use of CBD products. The FDA has issued numerous letters warning manufacturers of CBD products about false advertising and/or illegal marketing of CBD for unapproved uses to treat disorders such as Alzheimer's disease. In addition, prior evaluations of products containing CBD found that 69% were mislabeled in regards to the contents provided on the product labels. Given these matters, it is our intent to evaluate the efficacy of a topical CBD (TC) preparation in improving clinical outcomes in patients with chronic musculoskeletal joint pain. Specifically the investigators wish to establish the efficacy of TC, a product specifically formulated for topical application at pre-defined dosages.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of chronic musculoskeletal joint pain (arthritis, traumatic arthritis, osteoarthritis)
2. Adults ages 18 and over.
3. Medically stable without significant medical illness that would preclude treatment with either pharmacologic agent.
4. Have a safe, stable, living environment.

Exclusion Criteria

1. Unable to consent for research project.
2. Individuals less than 18 years of age.
3. Individuals with rheumatoid or other autoimmune types of arthritis.
4. Individuals diagnosed with SUD especially cannabis, as this may confound results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change in PGI-S | Two time points, before treatment and after 4 weeks.
  Patient Global Impression of Severity Scale from 1 to 7 with higher scores indicating worse condition
Change in PGI-C | Two time points, before treatment and after 4 weeks.
  Patient Global Impression of Change Scale from 1 to 7 with higher scores indicating worse condition
Change in QOLS | Two time points, before treatment and after 4 weeks.
  Quality of Life Scale Scale from 16 to 112, with higher scores indicating better condition

IPD SHARING:
Plan to Share IPD: No